CLINICAL TRIAL: NCT01507480
Title: The ELLIPSE Study: A Phase-1 Study Evaluating the Tolerance of Bevacizumab Nasal Spray to Treat Epistaxis in Hereditary Hemorrhagic Telangiectasia.
Acronym: ELLIPSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-650
Record Dates: First submitted 2011-12-06; First posted 2012-01-11 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2011-12

CONDITIONS: Rendu Osler Disease; Telangiectasia, Hereditary Hemorrhagic
Keywords: Hereditary Hemorrhagic Telangiectasia (HHT); Antiangiogenic therapies; Bevacizumab
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): This study is to be carried out sequentially (dose escalation) on 5 groups of 8 patients. Each group is made up of 6 verum and 2 placebos.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — There are five increasing doses of bevacizumab nasal spray (25mg/mL): 10 mg, 25 mg, 50 mg, 75, mg and 100 mg. Each test dose is a single dose divided into five fractions and administered into each nostril every 30 minutes for 2 hours:
  Other Names: AVASTIN

SUMMARY:
Antiangiogenic drugs, such as bevacizumab, are a new treatment strategy in Hereditary Hemorrhagic Telangiectasia (HHT). Its systemic administration in patients with HHT improves liver damage-related symptoms and epistaxis (cases reported and on-going study-ClinicalTrials.gov Identifier #NCT00843440-). To limit the systemic adverse effects of bevacizumab and to ease administration, a local administration seems suitable.

A clinical case recently showed the benefits of bevacizumab nasal spray in these patients. Its results were confirmed in a characterization study on bevacizumab transport through porcine nasal mucosa (in press).

It seems necessary to assess the tolerance and efficacy of bevacizumab nasal spray in humans for the treatment of epistaxis in HHT with a prospective phase 1 study.

The primary objective of the study is to evaluate the tolerance of increasing doses of bevacizumab administered as a nasal spray in patients with HHT-related epistaxis.

This phase-1, randomized, double-blind, placebo-controlled, monocentric study is to be carried out sequentially (dose escalation) on 5 groups of 8 patients. Each group is made up of 6 verum and 2 placebos.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who give voluntary, informed consent and sign a consent form.
* Patients affiliated with the French universal health care system.
* Patients treated for HHT, that has been confirmed clinically (presence of at lease 3 Curaçao criteria) and/or by molecular biology.
* Patients who fill out epistaxis tally sheets completely in the three months before inclusion.
* Patients who present severe epistaxis averaging over 30 minutes in the three months before inclusion ((duration M1 + duration M2 + duration M3) / 3).
* Patients whose number of red blood cell transfusions in the six months before inclusion is known.
* Patients who have not undergone nasal surgery in the three months before inclusion.

Exclusion Criteria:

* Pregnant women or women who could become pregnant during the study.
* Patients not affiliated with the French universal health care system.
* Patients who are protected adults according to the terms of the law (French public health laws).
* Refusal to give consent.
* Patients whose HHT diagnosis has not be confirmed clinically and/or by molecular biology.
* Infectious episode.
* Patients presenting unchecked hypertension at the time of inclusion (systolic BP > 150 mmHg and/or diastolic BP > 100 mmHg) with or without treatment. -Patients with hypertension can be included, once blood pressure levels have been controlled by appropriate medical treatment.
* Participation in another therapeutic trial in the 28 days before inclusion. Patients who have already being treated with bevacizumab by intravenous infusion.
* A known hypersensitivity to the active substance or one of its excipients.A known hypersensitivity to products containing Chinese hamster ovarian (CHO) cells or to other human or humanized recombinant antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tolerance | 3 months
  Evaluate the tolerance of increasing doses of bevacizumab administered as a nasal spray in patients with HHT-related epistaxis.

SECONDARY OUTCOMES:
Systemic passage and pharmacokinetics | 3 months
  Study the systemic passage and pharmacokinetics of bevacizumab in these patients.
Efficacy | 3 months
  Evaluate the efficacy of bevacizumab nasal spray on the appearance of epistaxis (number, frequency)
Efficacy | 3 months
  Evaluate the efficacy of bevacizumab nasal spray on hemoglobinema and ferritin
Efficacy | 3 months
  Evaluate the efficacy of bevacizumab nasal spray on the number of red blood cell transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Frederic FAURE, MD, Principal Investigator — Hospices Civils de Lyon

REFERENCES:
- [Derived] Dupuis-Girod S, Ambrun A, Decullier E, Samson G, Roux A, Fargeton AE, Rioufol C, Schwiertz V, Disant F, Chapuis F, Donazzolo Y, Paintaud G, Edery P, Faure F. ELLIPSE Study: a Phase 1 study evaluating the tolerance of bevacizumab nasal spray in the treatment of epistaxis in hereditary hemorrhagic telangiectasia. MAbs. 2014 May-Jun;6(3):794-9. doi: 10.4161/mabs.28025. Epub 2014 Jan 30. PMID 24481211
- See also: Related Info — http://www.rendu-osler.fr